CLINICAL TRIAL: NCT00821899
Title: Regeneration of Insulin Production in Patients With Type 1 Diabetes by Autologous Bone Marrow Blood Infusion
Brief Title: Bone Marrow Autotransplantation in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Enric Esmatjes, MD, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMATxDM1
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes type 1; bone marrow transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: administration of autologous bone marrow blood — administration of autologous bone marrow blood through magna pancreatic artery after femoral catheterization once during 12-month study period

SUMMARY:
This project evaluates the effectiveness of the administration of autologous bone marrow blood in patients with brittle type 1 diabetes mellitus to restore insulin secretion. After mobilization of hematopoietic progenitors (G-CSF) during 3 days, 50 to 90 mL of bone marrow blood will be obtained by multifunction in the posterior iliac crest. The material obtained will be implanted into the pancreas through the magna pancreatic artery after femoral catheterization.

ELIGIBILITY:
Inclusion Criteria:

* diabetes type 1 patients
* 18 to 50 years of age
* more than 5 years of evolution of the disease
* brittle diabetes (HbA1c > 8.5 % with intensified treatment or severe hypoglycemia episodes

Exclusion Criteria:

* history of cancer
* hematologic alterations
* infectious disease positivity (HIV, HCV etc.)
* diabetic nephropathy
* cardiac failure
* liver disease
* autoimmune systemic disease
* allergy to iodine contrast or anesthesia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Evaluate glycosylated hemoglobin 1,3,6, and 12 months after autologous bone marrow blood administration. | 12 months

SECONDARY OUTCOMES:
Evaluate number of hypoglycemias 1,3,6, and 12 months after autologous bone marrow blood administration. | 12 months
Evaluate insulin dose 1,3,6, and 12 months after autologous bone marrow blood administration. | 12 months
Evaluate GADab titers and treatment tolerance 1,3,6, and 12 months after autologous bone marrow blood administration. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Esmatjes Enric, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Enric Esmatjes, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona

REFERENCES:
- [Derived] Esmatjes E, Montana X, Real MI, Blanco J, Conget I, Casamitjana R, Rovira M, Gomis R, Marin P. Regeneration of insulin production by autologous bone marrow blood autotransplantation in patients with type 1 diabetes. Diabetologia. 2010 Apr;53(4):786-9. doi: 10.1007/s00125-010-1660-9. Epub 2010 Jan 26. No abstract available. PMID 20101385